CLINICAL TRIAL: NCT06312033
Title: Estradiol's Effect on Brain Volume and Connectivity in Naturally Cycling Women
Brief Title: Estradiol's Effect on Brain Volume and Connectivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Research Training Group 2804 (Other)
Collaborators: University Hospital Tübingen (Unknown); German Research Foundation (Other); Werner Reichardt Centrum für Integrative Neurowissenschaften (CIN) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: MRTG_P01
Record Dates: First submitted 2024-02-06; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Emotion Regulation; Estradiol
Keywords: brain structure; functional connectivity; sex hormones; women's mental health
MeSH Terms: conditions — Emotional Regulation | interventions — Estradiol

STUDY DESIGN:
Intervention Model Description: The intervention assessed the effect of estradiol administration on stress reactivity using a double blind randomized within -between placebo-controled design with repeated measures.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Neither participant or investigator knew the timepoint of drug or placebo administration. Pills were prepared by independent members of the university hospital.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- naturally cycling women starting with placebo (Experimental): naturally cycling women during early follicular phase starting with placebo (order was randomly selected)
  Interventions: Drug: Estradiol Valerate; Drug: Placebo
- naturally cycling women starting with estradiol (Experimental): naturally cycling women during early follicular phase starting with estradiol (order was randomly selected)
  Interventions: Drug: Estradiol Valerate; Drug: Placebo

INTERVENTIONS:
Drug: Estradiol Valerate — To elevate estradiol levels each woman has received 6mg on two consecutive days (total 12mg) of estradiol valerate (Progynova21©)
  Other Names: Progynova21
Drug: Placebo — Placebo (blue-colored hard gelatine capsules completely filled with a mixture of 99.5% mannitol and 0.5% Aerosil (fumed silica)) has been administered (placebo-controlled condition)

SUMMARY:
Ovarian hormones are not only modulators of cognitive function, emotion regulation and mental health, but also seem to affect brain plasticity and functional connectivity, During the menstrual cycle, women experience cyclic fluctuation of the ovarian hormone estradiol, which is closely associated with neuroplasticity/changes in brain structure in regions with high estradiol receptor density, such as the amygdala, hippocampus/parahippocampus, anterior cingulate cortex (ACC), striatum, and prefrontal cortex (PFC). Further functional connectivity between these areas seems to be associated with hormonal changes dependent on the menstrual cycle phase. But next to estradiol, also other hormones like progesterone fluctuate across the menstrual cycle. In the past, effects of ovarian hormone levels were often investigated in combination. However, one way to disentangle the impact of estradiol from that of other hormones on neuroplasticity, emotion regulation and mood states, can be the experimental increase of estradiol via estradiol administration. In this double-blinded within-subject study, women were administered either estradiol valerate or placebo during the early follicular phase (thus when ovarian hormone concentrations are low) before undergoing neuroimaging.

Parts of the study are already described in Rehbein et al., 2021 and 2022.

DETAILED DESCRIPTION:
In this project the investigators wanted to assess women with/without experimentally elevated estradiol (E2) levels in order to understand E2's effect on volume and resting state functional connectivity. Thus, women underwent fMRI (functional magnetic resonance imaging) scanning twice (with/without elevated E2) to deduce underlying neuronal activation. All participants underwent a structured assessment including demographical data, psychological/clinical data, e.g., structured clinical interview, anxiety traits, depression, emotion regulation traits, self-esteem as well as cognitive abilities, e.g., verbal intelligence, cognitive flexibility) and two (f)MRI measurements (T1/T2, separated by at least 2-3 months), including resting-state and anatomical scans as well as a behavioural emotion regulation task. At T1/T2 either E2 valerate or placebo was administered in a double-blinded, counterbalanced, randomized order.

E2 valerate administration: To experimentally elevate E2 concentrations each woman has received 6mg on two consecutive days (total 12mg) of E2 valerate (Progynova21©) Administration of E2 has been randomly distributed, so that women either received placebo (i.e. leading to an early follicular phase with low ovarian hormone levels) or E2 (i.e. leading to an early follicular phase with high E2 levels) first. Functional resting-state and anatomical data, emotion regulation performance, state anxiety, mood and depression scores have been acquired after the second pill intake. During the emotion regulation task women were asked to either (a) passively view aversive pictures or (b) down regulate their emotional response by e.g. changing their perspective on the picture and then rate their emotional state.

To assess changes in hormone concentrations (E2, progesterone, testosterone) blood samples were obtained before the first and after the second pill intake.

ELIGIBILITY:
Inclusion Criteria:

* Women, biologically female (assigned sex at birth)
* regular menstrual cycle lasting between 26 and 32 days
* right handedness

Exclusion Criteria:

* present or past mental, neurological or endocrine disorders
* use of hormonal contraceptives during the last six months
* any other medication intake,
* or past and present pregnancies
* Intake of antidepressants or neuroleptics
* contraindication for MRI

  * People with non-removable metal objects on or in the body
  * Tattoos (if not MRI-incompatible according to expert guidelines)
  * Pathological hearing or increased sensitivity to loud noises
  * Claustrophobia
  * Surgery less than three months ago
  * Neurological disease or injury
  * Moderate or severe head injury
  * Restricted vision

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Impact of E2 concentration on brain structure | From first measurement up to 6 months, with at least two months apart; each time: approx. 6 minutes during neuroimaging
  Brain structure (assessed via anatomical MRI scans, MPRAGE) will be compared between E2 and placebo conditions in regions of interest (ROI) (including amygdala, hippocampus/parahippocampus, ACC, striatum, and PFC).
Impact of E2 concentration and state emotion regulation on brain structure | From first measurement up to 6 months, with at least two months apart; each time: approx. 6 minutes during neuroimaging (structure) and 20 minutes (emotion regulation task)
  Brain structure (assessed via anatomical MRI scans, MPRAGE, in cm³) will be compared between E2 and placebo conditions in dependence of state emotion regulation ratings in ROIs (as above). State emotion regulation ratings obtained via the emotion regulation task (subjective rating ranging from -200 to 200).
Impact of E2 concentration and emotion regulation traits on brain structure | From first measurement up to 6 months, with at least two months apart; each time: approx. 6 minutes during neuroimaging
  Brain structure (assessed via anatomical MRI scans) will be compared between E2 and placebo conditions in dependence of emotion regulation traits in ROIs (as above). Emotion regulation traits assessed via the Heidelberg Form of Emotion Regulation (HFERST, ranging from 1 to 5) and the Emotion Regulation Questionnaire (ERQ, likert scale 1-7).
Impact of E2 concentration on resting state functional connectivity | From first measurement up to 6 months, with at least two months apart; each time: approx. 7 minutes during neuroimaging
  Resting state functional connectivity (assessed via resting state fMRI) will be compared between E2 and placebo condition in the whole brain and ROIs (as above).
Impact of E2 concentration and state emotion regulation on connectivity | From first measurement up to 6 months, with at least two months apart; each time: approx. 7 minutes (connectivity) and 20 minutes (emotion regulation task)
  Resting state functional connectivity (assessed via resting state fMRI) will be compared between E2 and placebo conditions in dependence of emotion regulation ratings in ROIs (as above). State emotion regulation ratings obtained via the emotion regulation task (subjective rating ranging from -200 to 200).
Impact of E2 concentration and emotion regulation traits on functional connectivity | From first measurement up to 6 months, with at least two months apart; each time: approx. 7 minutes (connectivity) during neuroimaging
  Resting state functional connectivity (assessed via resting state fMRI) will be compared between E2 and placebo conditions in dependence of emotion regulation traits in ROIs (as above). Emotion regulation traits assessed via the Heidelberg Form of Emotion Regulation (HFERST, ranging from 1 to 5) and the Emotion Regulation Questionnaire (ERQ, likert scale 1-7).
Impact of E2 concentration and associated structural brain changes on connectivity | From first measurement up to 6 months, with at least two months apart; each time before and after pill intake (6 minutes structure and 7 minutes connectivity)
  In order to investigate to which degree structural changes in association with E2 concentrations are related to changes in connectivity, both structure and connectivity were assessed via anatomical (MPRAGE) and resting state MRI scans.

SECONDARY OUTCOMES:
Impact of E2 concentration and self-esteem on brain structure | From first measurement up to 6 months, with at least two months apart; each time: approx. 6 minutes during neuroimaging
  Brain structure (assessed via anatomical MRI scans, MPRAGE) will be compared between E2 and placebo condition on dependence of self-esteem ratings in ROIs (as above). Self-esteem self-ratings assessed via the Rosenberg Self-Esteem Questionnaire (RSQ).
Impact of E2 concentration and self-esteem on functional connectivity | From first measurement up to 6 months, with at least two months apart; each time: approx. 7 minutes during neuroimaging
  Resting state functional connectivity (assessed via resting state fMRI) will be compared between E2 and placebo condition on dependence of self-esteem ratings in ROIs (as above). Self-esteem self-ratings assessed via the Rosenberg Self-Esteem Questionnaire (RSQ).
Impact of E2 concentration and subjective mood on brain structure | From first measurement up to 6 months, with at least two months apart; each time: approx. 6 minutes during neuroimaging
  Brain Structure (assessed via anatomical MRI scans, MPRAGE) will be compared between E2 and placebo condition in dependence of subjective mood in ROIs (as above). Ratings of subjective mood/affect obtained on the neuroimaging day.
Impact of E2 concentration and state anxiety on brain structure | From first measurement up to 6 months, with at least two months apart; each time: approx. 6 minutes during neuroimaging
  Brain Structure (assessed via anatomical MRI scans, MPRAGE) will be compared between E2 and placebo condition in dependence of state anxiety in ROIs (as above). Ratings of state anxiety (State Anxiety Inventory) obtained on the neuroimaging day
Impact of E2 concentration and subjective mood on functional connectivity | From first measurement up to 6 months, with at least two months apart; each time: approx. 7 minutes during neuroimaging
  Resting state functional connectivity (assessed via resting state MRI) will be compared between E2 and placebo condition in dependence of subjective mood in ROIs (as above). Ratings of subjective mood/affect obtained on the neuroimaging day.
Impact of E2 concentration and state anxiety on functional connectivity | From first measurement up to 6 months, with at least two months apart; each time: approx. 7 minutes during neuroimaging
  Resting state functional connectivity (assessed via resting state MRI) will be compared between E2 and placebo condition in dependence of state anxiety in ROIs (as above). Ratings of state anxiety (State Anxiety Inventory) obtained on the neuroimaging day.
Impact of E2 administration on E2 concentrations | From first measurement up to 6 months, with at least two months apart; each time before and after pill intake
  Changes in E2 concentrations(pmol/L), will be assessed from blood samples before and after pill intake.
Impact of E2 administration on E2-progesterone ratio | From first measurement up to 6 months, with at least two months apart; each time before and after pill intake
  Changes in E2-progesterone ratio will be assessed from blood samples before and after pill intake.
Impact of E2 administration on testosterone and progesterone concentration | From first measurement up to 6 months, with at least two months apart; each time before and after pill intake
  Changes in testosterone and progesterone concentrations (nmol/L) will be assessed from blood samples before and after pill intake.

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Derntl, Prof., Principal Investigator — Departement of Psychiatry & Psychotherapy
Locations (1):
- University of Tuebingen; Department of Psychiatry & Psychotherapy, Tübingen, Baden-Wurttemberg, Germany